CLINICAL TRIAL: NCT03520400
Title: PCI Alternative Using Sustained Exercise (PAUSE)
Brief Title: PCI Alternative Using Sustained Exercise
Acronym: PAUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F7374-R
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Percutaneous Intervention; coronary artery disease; exercise therapy
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease | interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Intervention Group (Experimental): Group receives one year of exercise and lifestyle intervention
  Interventions: Behavioral: Exercise Therapy
- PCI group (usual care) (No Intervention): Group receives standard clinical care with no intervention

INTERVENTIONS:
Behavioral: Exercise Therapy — Patients will adhere to one year of exercise therapy for the investigators' study. At minimum, subjects will aim to participate in approximately 30-60 minutes of aerobic exercise 5-7 days per week and 15-30 minutes of resistance/anaerobic exercise 2-3 times per week.
  Other Names: Exercise Training
  Arms: Exercise Intervention Group

SUMMARY:
Cardiovascular disease remains the leading cause of morbidity and mortality in the U.S. and is a major cause of disability in Veterans. Most of these deaths are due to coronary artery disease (CAD). The most common treatment for CAD is revascularization, an invasive procedure which usually involves placing a stent inside an artery that is diseased. However, exercise training is often overlooked because clinicians tend to focus on repairing the coronary circulation and the potential need for revascularization. Studies have shown that exercise training can be effective for patients with CAD and that it saves costs. In this study, invasive revascularization will be compared to a structured program of exercise training over one year. Comparisons will be made between groups for symptoms, coronary artery size and function using PET/CTA, and health care cost utilization.

DETAILED DESCRIPTION:
Despite advances in treatment options for cardiovascular disease (CVD), this condition remains the leading cause of morbidity and mortality in the U.S. and is a major cause of disability in Veterans. Percutaneous coronary intervention (PCI) is the treatment most often used in patients with various manifestations of coronary artery disease (CAD). While it is commonly assumed that PCI also reduces mortality, randomized trials have shown that PCI has no effect on mortality except in patients being treated for acute myocardial infarction. Over the last decade, the use of PCI has increased exponentially; between 1996 and 2007, the number of PCIs performed in the US has increased more than 4-fold, from approximately 300,000 to more than 1.3 million yearly. During this time, PCI has accounted for 10% of the overall increase in Medicare expenditures. In light of the extraordinary increase in the use of this technology in recent years, questions have been raised regarding the cost-effectiveness of PCI, the extent to which PCI is overused, and whether selected patients may benefit from optimal medical therapy in lieu of PCI. Cost analyses have suggested that the current rate of increase in PCI with DES is unsustainable for the U.S. healthcare system. Given the costs associated with PCI, there have been recent efforts to compare outcomes and effectiveness of PCI against non-invasive therapy.

There is a need to evaluate more judicious use of PCI, and to consider less costly interventions for at least some of the >1.3 million patients in the U.S. who undergo this procedure. Lifestyle intervention, including exercise training, is one option that has been shown to result in reduced symptoms, better exercise tolerance, improved quality of life and lower mortality. A growing body of data has demonstrated that exercise intervention improves coronary anatomy and lessens ischemia through enhanced endothelial function. While a significant proportion of health care expenditures are devoted to PCI and other invasive interventions for CVD, few health care resources are directed toward primary or secondary prevention. Recent studies have demonstrated that programs of cardiac rehabilitation, with and without implementation of intensive risk reduction, are cost effective. In part because of the financial interests associated with PCI, exercise and lifestyle intervention is rarely considered as a clinical treatment option in PCI candidates. A gap exists between the standard clinical treatment for CAD and the potential for non-invasive, less expensive and potentially more effective treatments for these patients. Previous efforts to quantify the effects of exercise and lifestyle intervention on coronary artery perfusion and anatomy have been limited to standard angiography. In recent years, improved technologies for imaging coronary perfusion and anatomy have been developed, which could provide important insights into the effects of exercise training on the heart. These include the combination of positron emission tomography and ultra-fast computed tomography angiography (CTA), commonly termed PET/CTA. PET provides information on the functional significance of anatomic stenoses by measuring myocardial blood flow and myocardial perfusion reserve. PET can also be used to evaluate coronary endothelial function by measurements of changes in myocardial blood flow in response to physical stimuli (i.e., cold pressor testing). The combination of CTA with PET also allows for improved attenuation correction. CTA, on the other hand, can noninvasively image the coronary arteries to determine the severity of stenosis and the amount of calcified and noncalcified plaque burden.

The investigators have termed the current proposal "PCI Alternative Using Sustained Exercise" (PAUSE) to reflect the potential for exercise training and lifestyle intervention as alternative therapies in selected PCI candidates.

Primary aim: To determine whether subjects with lesions amenable to PCI randomized to a 1 year exercise program and lifestyle intervention have greater improvement in coronary perfusion and function than those randomized to PCI.

Secondary analyses: The investigators will compare exercise test responses, health care costs, quality of life, and clinical outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients who have lesions appropriate for PCI based on American Heart Association/American College of Cardiology criteria will be considered for the study.
* Only patients with a good prognosis (annual mortality <2% based on VA multivariate scores (57, 58) will be considered.

Exclusion Criteria:

* Patients with left main disease or proximal LAD disease, or:

  * Unstable angina
  * A history of left ventricular dysfunction (EF 30%)
  * Pacemakers
  * Atrial fibrillation
  * Myocardial infarction within the last 3 months
  * Diabetes
  * Orthopedic problems interfering with the ability to exercise regularly

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Myers, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, de-identified data will be made available to collaborative institutions with whom the investigators are in contact.
Time Frame: Data collected will be available for 5 years after completion of the study.
Access Criteria: Following completion of the study in October 2018, the data will be available for 5 years.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Intervention Group | PCI Group (Usual Care)
Started | 37 | 14
Completed | 22 | 7
Not Completed | 15 | 7
Not completed — Physician Decision | 15 | 7

BASELINE CHARACTERISTICS:
Population: Subjects with suspected coronary artery disease undergoing percutaneous coronary intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention Group | PCI Group (Usual Care) | Total
Number analyzed (Participants) | 22 | 7 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 9
  >=65 years | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (3.8) | 69.0 (7.3) | 67.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 7 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 3 | 1 | 4
  White | 12 | 4 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion Reserve
Description: Measurement of myocardial blood flow has only been analyzed at baseline at this time. Intravenous 13NH3 will be used as the flow tracer and serial imaging with PET will be performed. Measurements will be performed at baseline, and after pharmacologic stress with dipyridamole. Myocardial blood flow at rest and following dipyridamole infusion will be expressed as ml flow/100 g/min. The myocardial perfusion reserve will be calculated as the ratio of the myocardial blood flow during stress (e.g. after dipyridamole) and the myocardial blood flow at rest. Commercially available software (Emory tool box) will be used to quantitatively analyze PET myocardial perfusion images.
Time Frame: baseline and 1 year
Population: Patients undergoing angiography for detection of coronary artery disease.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Exercise Intervention Group | PCI Group (Usual Care)
Number analyzed (Participants) | 22 | 7
Ratio
  Baseline | 2.76 (0.61) | 2.47 (0.48)
  1-year | 2.82 (0.56) | 2.52 (0.43)

2. Secondary Outcome: Peak VO2
Description: Peak VO2 will be determined at baseline and 1 year on a treadmill using an individualized ramp protocol with collection of continuous ventilatory gas exchange responses.
Time Frame: baseline and after 1 year
Population: Subjects undergoing angiography for detection of coronary artery disease.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Exercise Intervention Group | PCI Group (Usual Care)
Number analyzed (Participants) | 22 | 7
ml/kg/min
  Baseline | 20.21 (3.76) | 19.85 (6.5)
  1 Year | 22.4 (4.10) | 18.91 (5.92)

ADVERSE EVENTS:
Time Frame: 1-year
Arm/Group | Exercise Intervention Group | PCI Group (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/14
Other Adverse Events (participants affected / at risk) | 0/37 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-11-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03520400/Prot_SAP_000.pdf